CLINICAL TRIAL: NCT03090789
Title: Clinical Outcome Measures in Friedreich's Ataxia
Brief Title: FA Clinical Outcome Measures
Acronym: FA-COMS
Status: Active, not recruiting | Type: Observational
Sponsor: Friedreich's Ataxia Research Alliance (Other)
Collaborators: University of Rochester (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 01-002609
Record Dates: First submitted 2017-03-10; First posted 2017-03-27 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Friedreich Ataxia; Neuro-Degenerative Disease
Keywords: Friedreich Ataxia; Neuro-degenerative disease
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Biospecimen Retention: Samples With DNA — Optional sample collection offered to study participants; whole blood and/or cheek swab may be collected as a one-time procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Participant: Study participants can be individuals with either a clinical diagnosis or genetic confirmation of Friedreich ataxia. In addition, this study enrolls Friedreich ataxia carriers and unaffected controls.

SUMMARY:
This multicenter natural history study aims to expand the network of clinical research centers in FA, and to provide a framework for facilitating therapeutic interventions. In addition, this study will lead to the development of valid yet sensitive clinical measures crucial to outcome assessment of patients with Friedreich's Ataxia. This study will support genetic modifier studies, biomarker studies, and frataxin protein level assessments by building a sample repository.

This natural history study is no longer recruiting under this protocol NCT03090789 but remains actively recruiting under the harmonized study (UNIFAI) NCT06016946.

DETAILED DESCRIPTION:
Friedreich's ataxia (FA) is a rare autosomal recessive degenerative disorder characterized by ataxia, dysarthria, sensory loss, diabetes and cardiomyopathy. The discovery of the abnormal gene in FA and its product (frataxin) has provided insight into possible pathophysiological mechanisms and novel approaches to treatments in this disease. While such methods for assessing disease progression may be useful, evaluation in clinical trials will require specific clinical outcome measures.

This is a multicenter natural history study which aims to expand the network of clinical research centers specializing in Friedreich's Ataxia and to advance clinical care, research and therapeutic approaches in FA through the development and validation of clinical outcome measures. Study sites aim to collect quantitative serial clinical data on patients with FA and expand the existing research network. In addition, the study will support various genetic modifier studies, biomarker studies, and frataxin protein level assessments in patients with FA, in carriers, and in controls.

This study will recruit up to 2000 patients with Friedreich ataxia worldwide, to be assessed annually for up to 15 years. All individuals with a genetic or clinical diagnosis of FA can participate.

Study participation involves yearly assessments of a core set of clinical measures and quality of life assessment measures in addition to optional collection of a cheek swab and/or blood sample.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 4 to 80 years.
2. Genetically confirmed diagnosis of FA (for carrier/control cheek swab and blood samples this is not required).
3. Clinically confirmed diagnosis of FA, pending confirmatory genetic testing through a commercial or research laboratory (for carrier/control cheek swab and blood samples this is not required).
4. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1) Signs or symptoms of severe cardiomyopathy (such as congestive heart failure)

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with either a clinical diagnosis or genetic test confirmation of Friedreich ataxia. Study also accepts carriers of Friedreich ataxia along with healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2001-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Friedreich Ataxia Rating Scale | once every 1 year
  rating scale based on clinical neurologic examination

SECONDARY OUTCOMES:
9-hole peg test | once every 1 year
  timed test of fine motor skills performed as a set of four trials (two trials per hand), for patients with FA who are able to complete this testing
timed 25 foot walk | once every 1 year
  timed 25 foot walk is performed twice for patients with FA who are able to complete this testing. Assistive devices such as canes, service dogs, walkers, or crutches are permitted.
Vision assessment | once every 1 year
  High and low contrast visual acuity tested on patients with FA who are able to perform this test. Glasses or contact lenses are permitted.
Quality of Life Questionnaires | once every 1 year
  a set of quality of life questionnaires is administered for study participants with Friedreich ataxia. Questionnaires include items such as activities of daily living, overall opinion on health and function, and fatigue-related questions.

OTHER OUTCOMES:
Optional sample collection | once every 1 year
  study participants will be asked to provide a cheek swab and/or blood sample for a variety of different measures including frataxin protein level assessments or other biomarker tests

CONTACTS AND LOCATIONS:
Overall Officials: David Lynch, MD PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (14):
- United States (9):
  - UCLA Ataxia Center, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - University of Florida - Neurology, Gainesville, Florida
  - USF Ataxia Research Center, Tampa, Florida
  - Emory University Hospital - Neurology, Atlanta, Georgia
  - University of Iowa, Stead Family Children's Hospital, Iowa City, Iowa
  - Ohio State University - Neurology, Columbus, Ohio
  - Children's Hospital of Philadelphia - Neurology, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- Murdoch Childrens Research Institute, Parkville, Victoria, Australia
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
- All India Institute of Medical Sciences (Aiims), New Delhi, India
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No